CLINICAL TRIAL: NCT06477211
Title: A Multicenter Retrospective Study Identifying DNA 5mC Predictors for LUAD Prognosis
Brief Title: DNA Methylation Biomarkers to Predict Survival After Surgery for Lung Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Nanjing University (Other)
Collaborators: Peking Union Medical College Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Chen Qihan, Research Assistant, Nanjing University
Other Study IDs: Nanjing University
Record Dates: First submitted 2024-06-19; First posted 2024-06-27 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lung Adenocarcinoma; Surgery; Prognostic Cancer Model
Keywords: DNA methylation; prognosis; LUAD
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PUMCH: LUAD patients who underwent surgical treatment and were followed up at Peking Union Medical College Hospital
- NDTH: LUAD patients who received surgical treatment and were followed up at Nanjing Drum Tower Hospital

SUMMARY:
This study is designed to assess DNA 5-methylcytosine (5mC) methylation modifications in lung adenocarcinoma (LUAD) samples and develop a prognosis-predictive model for LUAD based on cancer tissue DNA 5mC levels. The research will link post-surgical recurrence and survival outcomes to the DNA 5mC profiles of patients. By collaborating with two hospitals in China, this multicentral study will utilize over three years of prognostic data from LUAD patients to validate the model's accuracy. Additionally, the research aims to explore the potential of the model in guiding adjuvant treatment strategies by comparing the differences in outcomes between high-risk patients who receive further treatment and those who do not. This study aspires to enhance future treatment planning for LUAD patients, providing personalized and effective therapeutic options based on precise prognostic predictions.

DETAILED DESCRIPTION:
* Model Development

  * The methylation data will be analyzed to identify specific 5mC methylation patterns associated with post-surgical recurrence and survival outcomes.
  * A prognostic model will be developed based on these methylation profiles to predict LUAD prognosis.
* Model Validation

  * Clinical data from LUAD patients at two hospitals in China, including over three years of follow-up information, will be used to validate the accuracy and reliability of the prognostic model.
  * Statistical methods will be applied to assess the model's predictive power and its ability to accurately stratify patients into different risk categories.
* Exploration of Follow-up and Adjuvant Therapy Guidance

  * The study will compare outcomes between high-risk patients who receive additional adjuvant treatment and those who do not, based on the risk categories identified by the prognostic model.
  * This comparison aims to explore the model's potential in guiding adjuvant therapy decisions, ultimately enhancing personalized treatment strategies and improving survival rates for LUAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed early-stage lung adenocarcinoma, or clinically diagnosed early-stage lung adenocarcinoma.
* Underwent surgical treatment
* Cancer tissues well paraffin-embedded or cryopreserved

Exclusion Criteria:

* Diagnosed with other serious illnesses
* Received other treatments before surgery
* Surgery to remove multiple cancerous tissues

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung adenocarcinoma patients
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Overall survival | 4years and/or 5years after surgery completion
  Subjects will be divided into high-risk and low-risk groups based on the DNA methylation model. The overall survival (OS) of these two groups will be compared to determine if there is a significant difference. Additionally, we will analyze whether there are significant differences in OS between high-risk and low-risk groups that received further treatment and those that did not.

SECONDARY OUTCOMES:
Disease-free survival | 4-year and/or 5-year after surgery completion
  Subjects will be divided into high-risk and low-risk groups based on the DNA methylation model. The disease-free survival (DFS) of these two groups will be compared to determine if there is a significant difference. Additionally, we will analyze whether there are significant differences in DFS between high-risk and low-risk groups that received further treatment and those that did not.

CONTACTS AND LOCATIONS:
Overall Officials: Qihan Chen, PhD, Principal Investigator — Nanjing University
Locations (1):
- Nanjing Drum Tower hospital, Nanjing, Jiangsu, China